CLINICAL TRIAL: NCT02283710
Title: The Effect of Pentoxifylline on Liver Function Tests in Non-alcoholic Fatty Liver Disease Patients Refereed to Sina Hospital Gastroenterology Clinic
Brief Title: The Effect of Pentoxifylline on Liver Function Tests in Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Raika Jamali, MD, Associate Professor of Medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9011160012
Record Dates: First submitted 2014-11-01; First posted 2014-11-05 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Fatty Liver
Keywords: Pentoxifylline; Aminotransferase; Steatohepatitis
MeSH Terms: conditions — Fatty Liver | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pentoxifylline + lifestyle modification (Experimental): Pentoxifylline for 6 months plus obtaining ideal body weight by calorie restriction diet and programmed physical activity.
  Interventions: Drug: Pentoxifylline; Behavioral: Lifestyle modification
- Lifestyle modification (Experimental): Obtaining ideal body weight by calorie restriction diet and programmed physical activity.
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline 600 mg BD
  Arms: Pentoxifylline + lifestyle modification
Behavioral: Lifestyle modification — obtaining ideal body weight by calorie restriction diet and programmed physical activity.

SUMMARY:
This randomized double blind clinical trial was performed in patients with non-alcoholic fatty liver disease.They were randomly assigned to lifestyle modification alone or lifestyle modification plus Pentoxifylline groups. Liver function tests, metabolic profile and anthropometric measurements were checked at baseline and six months later.

DETAILED DESCRIPTION:
This randomized double blind clinical trial was performed in patients with the evidence of fatty liver in ultrasonography. After excluding other causes, participants with persistent elevated serum aminotransferase levels were presumed to have NAFLD. Those with NAFLD liver fat score greater than (-0.64) were enrolled. They were randomly assigned to lifestyle modification alone or lifestyle modification plus Pentoxifylline groups. Fasting serum glucose, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, triglyceride, cholesterol, high and low-density lipoprotein,homeostasis model assessment-insulin resistance(HOMA-IR), and anthropometric measurements (body mass index and waist circumference) were checked at baseline and six months later.

ELIGIBILITY:
Inclusion Criteria:

Patients with persistent elevated aminotransferase levels and the evidence of fatty liver in ultrasonography, who were referred to a gastroenterology clinic.

Exclusion Criteria:

* alcohol use (more than 20 gram per day in men and 10 gram per day in women per day),
* heart disease (ischemic or congestive),
* hepatic disease (viral hepatitis, autoimmune hepatitis, wilson disease, hemochromatosis, liver mass lesion),
* renal disease (serum creatinine concentration of > 1.5 mg/dl),
* any severe systemic co-morbidities, neoplasm,
* using any hepatotoxic medication during the past 3 months,
* pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline serum alanine aminotransferase at 6 months | 6 months

SECONDARY OUTCOMES:
Change from baseline serum aspartate aminotransferase at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raika Jamali, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Gastroenterology clinic, Sina Hospital, Tehran, Tehran Province, Iran